CLINICAL TRIAL: NCT06075160
Title: Prospective Evaluation of Long-term Clinical Outcomes After Resting Full-cycle Ratio (RFR)-Guided Percutaneous Coronary Revascularization; A Multi-center, International, Single Arm Interventional, Comparing Registry (COMFORT Study)
Brief Title: Resting Full-cycle Ratio (RFR)-Guided Revascularization
Status: Recruiting | Type: Observational
Sponsor: Sejong General Hospital (Other)
Collaborators: Wonju Severance Christian Hospital (Other); Hospital San Carlos, Madrid (Other); Seoul St. Mary's Hospital (Other); Dong-A University Hospital (Other); Gyeongsang National University Hospital (Other); Soon Chun Hyang University (Other); Keimyung University Dongsan Medical Center (Other); Ulsan University Hospital (Other); Seoul National University Bundang Hospital (Other); Kosin University Gospel Hospital (Other); Pusan National University Hospital (Other)
Responsible Party: Principal Investigator, Hyun Jong Lee, MD, PhD, Sejong General Hospital
Other Study IDs: COMFORT Vesion 2.6
Record Dates: First submitted 2023-10-03; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Coronary Artery Disease
Keywords: physiologic assessment; intermediate stenosis
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Resting full-cycle ratio (RFR)-guided revascularization — The decision of coronary intervention is based on an RFR cut-value of 0.89. If RFR ≤ 0.89, target lesion will be revascularized, and if RFR > 0.89, PCI will be deferred. However, even if RFR ≤ 0.89, PCI can be deferred if the RFR gradient of the lesion ≤ 0.02, or if the diffused type of stenosis, because physiological gain is expected to be very low.
Diagnostic Test: Fractional flow ratio (FFR)-guided revascularization — Study participants of FFR-guided PCI arm will be selected from a large-scaled, ongoing FFR registry. The decision of coronary intervention is based on an FFR cut-value of 0.80. If FFR ≤ 0.80, target lesion will be revascularized, and if RFR > 0.80, PCI will be deferred.

SUMMARY:
The purpose of this study is to compare the clinical outcomes of a 2-year follow-up to determine whether RFR-guided coronary intervention is non-inferior to FFR-guided coronary intervention in patients with intermediate coronary stenosis.

DETAILED DESCRIPTION:
Myocardial ischemia is a key determinant of clinical prognosis in patients with coronary artery disease. In this regard, functional assessment of intermediate coronary stenoses with transtenotic pressure ratios provides a more accurate measure of stenosis-derived myocardial ischemia in comparison to conventional coronary angiography (3-5). One of the major clinical benefit of fractional flow reserve (FFR) is that, by acting as a gatekeeper, non-ischemia-causing lesions suitable for optimal medical treatment can be accurately identified, avoiding unnecessary coronary stenting. However, despite being support with the highest level of recommendation by the current guidelines for guiding clinical-decision making, adoption of FFR in the real world practice is still very low, mainly due to the need of hyperemic agents like adenosine that frequently cause patient discomfort, and time consumption. To overcome such limitations of pressure-wire derived index from the need of adenosine, other alternatives have been looking for over the last years. Instantaneous wave-free ratio (iFR), a resting trans-stenotic pressure index obtained as the ratio of distal coronary pressure to aortic pressure during the diastolic wave-free period, demonstrated a good diagnostic accuracy to define functional significance of coronary lesions without need of adenosine, using FFR as reference. Recently, two large, randomized trials demonstrated that iFR-guided coronary revascularization is clinically non-inferior to FFR-guided revascularization with respect to one-year risk of major adverse cardiac events. Accordingly, like FFR, iFR is now receiving the highest level of recommendations to guide clinical decision making in patients with stable intermediate coronary stenosis. A new adenosine-free index, the resting full-cycle ratio (RFR), has recently emerged. RFR is defined as the lowest ratio of intracoronary distal pressure to aortic pressure under resting condition, irrespective of systole or diastole, and has demonstrated equivalent diagnostic performance to iFR. RFR has an advantage over iFR, because it is not limited by sensitive land marking of components of the pressure waveform unlike iFR.

This novel physiologic index without the need of adenosine has the potential to increase the worldwide adoption of coronary physiology in guiding coronary revascularization in daily clinical practice. However, there is a paucity of important data regarding clinical outcomes of RFR-guided revascularization strategy. We hypothesize long-term clinical outcome of RFR-guided revascularization is non-inferior to that of FFR-guided revascularization, and it reduce the rate of PCI than FFR-guided revascularization. Therefore, we sought to investigate the long-term effectiveness and safety of RFR-based decision making in patients with one or more intermediate coronary stenosis, and to assess whether it is non-inferior to FFR-guided revascularization.

ELIGIBILITY:
Inclusion Criteria:

* Patients with intermediate coronary artery stenosis (visually 50-90% diameter stenosis) who decided to undergoing a RFR-guided coronary intervention according to clinical necessity
* Patients who voluntarily decided to participate in this study and signed informed consent

Exclusion Criteria:

* Severe left ventricular systolic dysfunction (LVEF <30%)
* Cardiogenic shock
* Culprit vessel in acute coronary syndrome
* Donor vessel to supply chronic total occlusion lesion of non-target vessel
* Symptomatic valvular heart disease or cardiomyopathy
* Hemodynamic instability at the time of intervention (heart rate <50 beats per minute, systolic blood pressure <90mmHg)
* Previous CABG with patent grafts to the interrogated vessel
* Pregnancy or breastfeeding
* Non-cardiac co-morbid conditions are present with life expectancy <1 year or that may result in protocol non-compliance

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with intermediate coronary artery stenosis, who need functional evaluation
Sampling Method: Non-Probability Sample
Enrollment: 1167 (Estimated)
Dates: Start 2022-07-27 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
A composite of death from any cause, non-fatal myocardial infarction, or unplanned revascularization | At 2-year

SECONDARY OUTCOMES:
Target lesion failure | At 2-year
  A composite of cardiac death, target vessel MI, or target lesion revascularization
Target vessel failure | At 2-year
  A composite of cardiac death, target vessel MI, or target vessel revascularization
Death from any cause | At 2-year
Cardiovascular death | At 2-year
Cardiac death or non-fatal MI | At 2-year
Non-fatal MI | At 2-year
Any unplanned revascularization | At 2-year
Target vessel revascularization | At 2-year
Target lesion revascularization | At 2-year

CONTACTS AND LOCATIONS:
Locations (1):
- Sejong general hospital, 91-121 Sosa 2-Dong, Sosa-Gu, Bucheon-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No